CLINICAL TRIAL: NCT03445650
Title: A Phase 3 Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Trial to Evaluate the Safety and Efficacy of ADX-102 1% Topical Dermal Cream (Reproxalap) in Subjects With Sjögren-Larsson Syndrome (SLS)
Brief Title: RESET Trial - Part 1 - A Phase 3 Trial in Subjects With Sjögren-Larsson Syndrome (SLS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-SLS-006
Record Dates: First submitted 2018-02-14; First posted 2018-02-26 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Sjogren-Larsson Syndrome
Keywords: ADX-102, Sjögren-Larsson Syndrome
MeSH Terms: conditions — Sjogren-Larsson Syndrome | interventions — reproxalap; Skin Cream

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADX-102 1% Topical Dermal Cream (reproxalap) (Experimental)
  Interventions: Drug: ADX-102 1% Topical Dermal Cream (reproxalap)
- Vehicle of ADX-102 Topical Dermal Cream (Placebo Comparator)
  Interventions: Drug: Vehicle of ADX-102 Topical Dermal Cream

INTERVENTIONS:
Drug: ADX-102 1% Topical Dermal Cream (reproxalap) — ADX-102 1% Topical Dermal Cream administered approximately every 24 hours for 6 months.
  Arms: ADX-102 1% Topical Dermal Cream (reproxalap)
Drug: Vehicle of ADX-102 Topical Dermal Cream — Vehicle of ADX-102 Topical Dermal Cream administered approximately every 24 hours for 6 months.
  Arms: Vehicle of ADX-102 Topical Dermal Cream

SUMMARY:
A Phase 3 Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Trial to Evaluate the Safety and Efficacy of ADX-102 1% Topical Dermal Cream in Subjects with Sjögren-Larsson Syndrome (SLS).

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged 3 years or older
* Subject has a genetically-confirmed diagnosis of SLS.
* Subject has active ichthyosis that is Grade 2 or higher on the Visual Index Ichthyosis Severity (VIIS) score.
* Females of child-bearing potential: Negative pregnancy test at Screening and Baseline Visits.

Exclusion Criteria:

* Subject has evidence of a serious active infection.
* Systemic or topical retinoids or other topical medications, not including emollients, within the past 30 days Baseline Visit 1.
* Subject has received an investigational systemic or topically administered drug within the past 30 days prior to Baseline Visit 1.
* Subject is currently receiving immunosuppressive therapy, including intermittent or low-dose systemic corticosteroids.
* Subject has a known allergic reaction to any ingredients of study drug formulation.
* Subject has any clinically significant laboratory test abnormalities or a history of any other condition that, in the opinion of the Investigator, could compromise the subject's ability to comply with the protocol or that could compromise the subject's safety or the interpretation of the study results.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ADX-102 1% Topical Dermal Cream: ADX-102 1% Topical Dermal Cream: ADX-102 1% Topical Dermal Cream administered approximately every 24 hours for 6 months in Part 1
- Vehicle Topical Dermal Cream: Vehicle Topical Dermal Cream: Vehicle of ADX-102 Topical Dermal Cream administered approximately every 24 hours for 6 months in Part 1
Period: Overall Study
Arm/Group | ADX-102 1% Topical Dermal Cream | Vehicle Topical Dermal Cream
Started | 7 | 4
Completed | 6 | 3
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADX-102 1% Topical Dermal Cream | Vehicle Topical Dermal Cream | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.1 (7.78) | 9.5 (6.35) | 15.0 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  White | 5 | 3 | 8
  Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 4 | 11
Height [Mean (Standard Deviation); unit: centimeters] | 150.38 (24.583) | 125.68 (29.287) | 141.39 (27.850)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 48.81 (18.708) | 29.18 (18.864) | 41.67 (20.367)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 20.5 (3.36) | 16.8 (2.89) | 19.1 (3.57)
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.4 (0.39) | 1.0 (0.42) | 1.3 (0.43)

OUTCOME MEASURES:

1. Primary Outcome: Visual Index Ichthyosis Severity (VIIS) Scaling Score as Assessed by the Investigator in ADX-102 Treated Patients
Description: Change from baseline using the Visual Index Ichthyosis Severity (VIIS) Scaling Score (0 = least, 4 = most), where a higher value represents a worse outcome, in ADX-102 treated patients
Time Frame: Efficacy assessment period (Week 1 through Week 24), where Baseline is Day 1.
Population: modified intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ADX-102 1% Topical Dermal Cream
Number analyzed (Participants) | 6
units on a scale | -0.7 (0.22)

ADVERSE EVENTS:
Time Frame: The period of time when adverse events were collected was approximately 28 weeks.
Arm/Group | ADX-102 1% Topical Dermal Cream | Vehicle Topical Dermal Cream
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 6/7 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADX-102 1% Topical Dermal Cream (N=7) | Vehicle Topical Dermal Cream (N=4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hordeolum (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Feeling hot (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 2 | 0
Ichthyosis (Congenital, familial and genetic disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Eosinophil count increased (Investigations) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03445650/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03445650/SAP_003.pdf